CLINICAL TRIAL: NCT05575050
Title: Impact of Teeth Brushing on Bacterial Microbiota and Healthcare-associated Infections in Ventilated COVID-19 Patients
Brief Title: Impact of Teeth Brushing in Ventilated COVID-19 Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital in Krakow (Other)
Responsible Party: Principal Investigator, Mateusz Fiema, MD, University Hospital in Krakow
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1072.6120.333.2020
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Microbial Colonization; COVID-19 Respiratory Infection; Dysbiosis; VAP - Ventilator Associated Pneumonia; HAI
Keywords: oral microbiota; healthcare-associated infection
MeSH Terms: conditions — Communicable Diseases; Dysbiosis; Pneumonia, Ventilator-Associated; Cross Infection | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Patients were divided into 2 groups depending on the oral care procedure:
  1. Standard oral procedure (cleaning and moisturizing of oral cavity, suction of excess fluid)
  2. Extended oral procedure (cleaning and moisturizing of oral cavity, teeth brushing, suction of excess fluid) The procedures were performed twice daily in each patient. The detailed information on these procedures is included in the Appendix 1. The allocation protocol was based on patients' location in the ward. Each room was assigned with one type procedure (standard- even number or extended - uneven number of room), that was permanent during the study period.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard oral procedure (Active Comparator): Standard mouth cleaning protocol (without brushing) included:
  1. Preparation of sterile catheter (12F lub 14F), suction of excess fluid from the oral cavity.
  2. Using Sage Suction Swab (Toothette®), soaking in Perox-A-Mint Solution and cleaning with circular movements of each mucosal site for 10 seconds:
     1. Right cheek mucosa and right upper quadrant
     2. Left cheek mucosa and left upper quadrant
     3. Left lower buccal quadrant
     4. Right lower buccal quadrant
  3. Moisturizing with Mouth Moisturizer /firma/ of oral cavity mucosa, tongue and lips.
  4. Repeated suction of excess fluid from the oral cavity.
  Interventions: Procedure: Oral Procedure
- Extended oral procedure (Active Comparator): Extended mouth cleaning protocol (with brushing) included:
  1. Preparation of sterile catheter (12F lub 14F), suction of excess fluid from the oral cavity.
  2. Teeth brushing (each teeth quadrant for 30) using Sage Untreated Suction Toothbrush (SUST) connected to suction unit, moistured with sterile water.
  3. Using Sage Untreated Suction Toothbrush (SUST) moisturised with sterile water and cleaning with circular movements of each mucosal site for 10 seconds:
     1. Right cheek mucosa and right upper quadrant
     2. Left cheek mucosa and left upper quadrant
     3. Left lower buccal quadrant
     4. Right lower buccal quadrant
  4. Moisturizing with Mouth Moisturizer of oral cavity mucosa, tongue and lips.
  5. Repeated suction of excess fluid from the oral cavity.
  Interventions: Procedure: Oral Procedure

INTERVENTIONS:
Procedure: Oral Procedure — Interventions included 2 variants of oral hygienic procedures. One was extended of teeth brushing.

SUMMARY:
The aims of this study were:

1. Observation of dynamics in oral microbiota and its association with the incidence of HAIs and VAP in mechanically ventilated COVID-19 patients in an ICU setting
2. Evaluation of the incidence of HAIs and VAP and their association with oral bacteriobiota in mechanically ventilated COVID-19 patients in an ICU setting
3. Assessment of impact of different oral hygienic procedures on oral microbiota, the incidence of HAI and patients' safety in mechanically ventilated COVID-19 patients in an ICU setting approaches to oral care in an ICU setting

Intervention of oral hygienic procedures implemented in study:

Patients were divided into 2 groups depending on the oral care procedure:

1. Standard oral procedure (cleaning and moisturizing of oral cavity, suction of excess fluid)
2. Extended oral procedure (cleaning and moisturizing of oral cavity, teeth brushing, suction of excess fluid)

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection confirmed by real-time reverse transcriptase-polymerase chain reaction (RT-PCR) assay of nasal and pharyngeal swabs upon hospital admission
* Signed consent to participate in the study
* Patients admitted to ICU
* Intubation due to COVID-19 related pneumonia and acute respiratory distress syndrome (ARDS) within 24 hours preceding study procedures

Exclusion Criteria:

* No consent to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Healthcare-associated infection | one month
  Healthcare-associated infection (HAI) incidence was measured.

SECONDARY OUTCOMES:
Oral cavity assessment | one month
  Using The Beck Oral Assessment Scale (BOAS)
Frequency of identification of Enterococcus fecalis, Acinetobacter baumannii, Klebsiella pneumoniae. | one month
  Frequency of identification of Enterococcus fecalis, Acinetobacter baumannii, Klebsiella pneumoniae in different samples from oral cavity taken from ventilated COVID-19 patients on Intensive Care Unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Hospital Kraków, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided